CLINICAL TRIAL: NCT06168331
Title: Chinese Community Inpatient Thromboembolism: a Cross-sectional Study
Brief Title: Chinese Community Inpatient Thromboembolism
Acronym: COMET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhi-chun Gu, associate professor of pharmacy, RenJi Hospital
Other Study IDs: IIT-2023-0216
Record Dates: First submitted 2023-10-31; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; Community hospitalization
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter cross-sectional study conducted at 20 centers. Data of existing inpatients in 20 community hospitals were collected. Information collected included demographic, co-morbidities, co-medication, laboratory tests, imaging tests, and anticoagulant use. Based on Caprini, Padua, Khorana and PAPT rating tables, VTE risk assessment was carried out for inpatients from 20 community hospitals, and VTE risk stratification of patients and prevention of high-risk VTE patients were analyzed. Blood samples of inpatients were collected to determine coagulation function indicators. VTE screening was performed on hospitalized patients using color Doppler ultrasound to determine the incidence of VTE in community hospitalized patients. On this basis, the predictive efficacy of different VTE risk scores on community hospitalized patients was compared, and a new VTE risk score conforming to community hospitalized patients was constructed.

DETAILED DESCRIPTION:
This study was a prospective, multicenter, observational cohort study conducted in a cross-section of 20 eligible community hospitals.

Data of existing inpatients in 20 community hospitals were collected. Information collected included demographic, co-morbidities, co-medication, laboratory tests, imaging tests, and anticoagulant use. Inpatients from 20 community hospitals were evaluated for VTE risk by integrating scores such as Caprini, Padua, Khorana and PAPT, and their ability to perform activities of daily living was also evaluated. The stratification of VTE risk and the prevention of VTE in high-risk patients were analyzed, and the efficacy of different VTE risk scores in predicting VTE in community inpatients was compared. VTE risk score was constructed by Delphi method to simplify the clinical VTE evaluation process.

Delphi method was used to construct a VTE risk scoring process: 1) This study initially proposed several VTE risk indicators such as age, length of stay and score of autonomous activity ability through literature review. After analysis, discussion and rectification, the research team members screened the indicators according to the construction principles of the indicator system, and finally preliminatively determined the level and quantity of sensitive indicators. 2) Design expert letter questionnaire: This study plans to conduct a total of 3 rounds of letter questionnaire, which will be distributed and recovered by face-to-face presentation or email. 15 clinical experts with senior titles who have worked in VTE related research fields for more than 10 years, including clinicians, clinical pharmacists and nurses, etc., will be invited. Experts will evaluate all levels and indicators one by one. Likert 5-level scoring method will be adopted for the importance score, and 1-5 points will be assigned according to "not important" to "very important". Modifications, additions or other comments on indicators will be recorded in the expert opinion column. 3) Pairwise comparison of indicators at all levels in the third round of expert letter questionnaire was carried out, and the pairwise comparative importance of each indicator was assigned by the 9-level scale of analytic Hierarchy Process (AHP). Matrix judgment and weight were determined according to the expert evaluation results. Determine the final VTE risk score.

Lower extremity venous ultrasound was performed on more than 1000 patients to obtain the current incidence of VTE among hospitalized patients in the community.

Blood samples were collected from more than 1000 patients, and blood samples from hospitalized patients were collected to determine coagulation function indexes, including prothrombin time, fibrinogen, partial thromboplastin time, thrombin time, fibrin degradation products, D-D dimer, and coagulation active factors.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in community service centers

  * Patients or guardians agree with the study plan and sign the informed consent.

Exclusion Criteria:

* Outpatients in community service centers

  * The patient or guardian does not agree to sign the informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inpatients from 20 community health service centers in Shanghai.
Sampling Method: Probability Sample
Enrollment: 1152 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower extremity venous ultrasound VTE event | This is a cross-sectional study， patients will be examined Day0 when incorporated into study
  Both lower limb venous B-ultrasonography will be performed on the patients to examine whether the patient has VTE event

SECONDARY OUTCOMES:
D-Dimer D-Dimer D-Dimer D-Dimer level | This is a cross-sectional study， patients will be examined Day0 when incorporated into study
  Indicators of coagulation function in patients, D-D dimer will be assayed to be the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy, Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided